CLINICAL TRIAL: NCT06612398
Title: Effect of a Preoperative Preparation Video on Preoperative Anxiety Among Children Undergoing Dental Treatment Under General Anesthesia
Brief Title: Effect of a Preparation Video on Preoperative Anxiety in Children Undergoing Dental Treatment Under GA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 72/149/2022
Record Dates: First submitted 2024-08-30; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-08

CONDITIONS: Preoperative Anxiety

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Research Assistant who evaluated patient's anxiety levels did not know who watched the intervention and who did not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Participants received the standard care provided upon arrival and being admitted to the hospital, involving only a verbal explanation of the anaesthesia induction process.
- Preoperative preparation video (Experimental): On the night before the surgery, participants were presented with an animated video illustrating the story of a child's journey through the hospital facilities, including the anaesthesia induction, and the postoperative return home.
  Interventions: Behavioral: Preoperative preparation video

INTERVENTIONS:
Behavioral: Preoperative preparation video — An animated video illustrating the story of a child's journey through the hospital facilities, including the anaesthesia induction, and the postoperative return home.
  Arms: Preoperative preparation video

SUMMARY:
The present study investigated the effect of an animated preoperative preparation video in mitigating preoperative anxiety among children receiving comprehensive dental treatment under General Anesthesia (GA).

DETAILED DESCRIPTION:
This randomised controlled trial, conducted at King Abdullah University Hospital (KAUH) over an eight-month period from February to October 2023, focused on children aged four to seven years undergoing comprehensive dental treatment under GA. Participants were randomly assigned to either the control group or the study group. Participants in the control group received the standard care provided upon arrival at the Day Case Unit (DCU) at KAUH, involving only a verbal explanation of the anaesthesia induction process. In contrast, on the night before the surgery, participants in the study group were presented with an animated video illustrating the story of a child's journey through the hospital facilities, including the anaesthesia induction, and the postoperative return home. Additionally, all parents watched the video alongside their children and provided positive comments on its content. The primary outcome assessed was the children's preoperative anxiety measured by modified Yale Preoperative Anxiety Scale (m-YPAS) and Visual Facial Anxiety Scale (VFAS), allowing for an evaluation of the intervention's impact.

ELIGIBILITY:
Inclusion Criteria:

* Children who are healthy, with American Society of Anesthesiologists (ASA) Grade 1 and 2 status.
* Age 4-7 years.
* Children undergoing GA for the first time who require comprehensive dental rehabilitation.

Exclusion Criteria:

* Presence of a systemic disease, as well as mental, cognitive, and intellectual disabilities.
* Presence of visual or auditory disability.
* Participants who refuse to answer subjective scales due to heightened anxiety levels.
* Participants with no access to internet services.
* Presence of active severe dental pain and/or facial abscess as it could affect the participant's state anxiety.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
modified Yale Preoperative Anxiety Scale | 1 day
  Observational anxiety scale, values (23.3-100) with higher scores indicating higher levels of anxiety
Visual Facial Anxiety Scale | 1 day
  Self-report anxiety scale, values (0-10) with higher scores indicating higher levels of anxiety

SECONDARY OUTCOMES:
Face, Legs, Activity, Cry, Consolability scale | 1 day
  Observational pain scale, values (0-10) with higher scores indicating higher levels of pain
Pediatric Anesthesia Emergence Delirium scale | 1 day
  Observational emergence delirium scale, values (0-20) with higher scores indicating higher levels of emergence delirium

CONTACTS AND LOCATIONS:
Overall Officials: Mawia Bataineh, Doctor, Study Chair — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995
- [Background] Al-Jundi SH, Mahmood AJ. Factors affecting preoperative anxiety in children undergoing general anaesthesia for dental rehabilitation. Eur Arch Paediatr Dent. 2010 Feb;11(1):32-7. doi: 10.1007/BF03262707. PMID 20129031
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Kim J, Chiesa N, Raazi M, Wright KD. A systematic review of technology-based preoperative preparation interventions for child and parent anxiety. Can J Anaesth. 2019 Aug;66(8):966-986. doi: 10.1007/s12630-019-01387-8. Epub 2019 May 16. PMID 31098960
- [Background] Schwartz BH, Albino JE, Tedesco LA. Effects of psychological preparation on children hospitalized for dental operations. J Pediatr. 1983 Apr;102(4):634-8. doi: 10.1016/s0022-3476(83)80211-x. PMID 6834205
- [Background] Wright KD, Raazi M, Walker KL. Internet-delivered, preoperative, preparation program (I-PPP): Development and examination of effectiveness. J Clin Anesth. 2017 Jun;39:45-52. doi: 10.1016/j.jclinane.2017.03.007. Epub 2017 Mar 27. PMID 28494907
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Cao X, Yumul R, Elvir Lazo OL, Friedman J, Durra O, Zhang X, White PF. A novel visual facial anxiety scale for assessing preoperative anxiety. PLoS One. 2017 Feb 14;12(2):e0171233. doi: 10.1371/journal.pone.0171233. eCollection 2017. PMID 28196099
- [Background] Crellin DJ, Harrison D, Santamaria N, Babl FE. Systematic review of the Face, Legs, Activity, Cry and Consolability scale for assessing pain in infants and children: is it reliable, valid, and feasible for use? Pain. 2015 Nov;156(11):2132-2151. doi: 10.1097/j.pain.0000000000000305. PMID 26207651
- [Background] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Background] Koo TK, Li MY. A Guideline of Selecting and Reporting Intraclass Correlation Coefficients for Reliability Research. J Chiropr Med. 2016 Jun;15(2):155-63. doi: 10.1016/j.jcm.2016.02.012. Epub 2016 Mar 31. PMID 27330520
- [Background] Powell R, Scott NW, Manyande A, Bruce J, Vogele C, Byrne-Davis LM, Unsworth M, Osmer C, Johnston M. Psychological preparation and postoperative outcomes for adults undergoing surgery under general anaesthesia. Cochrane Database Syst Rev. 2016 May 26;2016(5):CD008646. doi: 10.1002/14651858.CD008646.pub2. PMID 27228096
- [Background] Kain ZN, Caldwell-Andrews AA, Mayes LC, Weinberg ME, Wang SM, MacLaren JE, Blount RL. Family-centered preparation for surgery improves perioperative outcomes in children: a randomized controlled trial. Anesthesiology. 2007 Jan;106(1):65-74. doi: 10.1097/00000542-200701000-00013. PMID 17197846
- [Background] Rantala A, Pikkarainen M, Miettunen J, He HG, Polkki T. The effectiveness of web-based mobile health interventions in paediatric outpatient surgery: A systematic review and meta-analysis of randomized controlled trials. J Adv Nurs. 2020 Aug;76(8):1949-1960. doi: 10.1111/jan.14381. Epub 2020 Apr 22. PMID 32281673
- [Background] Demblon MC, Bicknell C, Aufegger L. Systematic review of the development and effectiveness of digital health information interventions, compared with usual care, in supporting patient preparation for paediatric hospital care, and the impact on their health outcomes. Front Health Serv. 2023 Apr 6;3:1103624. doi: 10.3389/frhs.2023.1103624. eCollection 2023. PMID 37089454
- [Background] Lee J, Lee J, Lim H, Son JS, Lee JR, Kim DC, Ko S. Cartoon distraction alleviates anxiety in children during induction of anesthesia. Anesth Analg. 2012 Nov;115(5):1168-73. doi: 10.1213/ANE.0b013e31824fb469. Epub 2012 Sep 25. PMID 23011563
- [Background] Eijlers R, Dierckx B, Staals LM, Berghmans JM, van der Schroeff MP, Strabbing EM, Wijnen RMH, Hillegers MHJ, Legerstee JS, Utens EMWJ. Virtual reality exposure before elective day care surgery to reduce anxiety and pain in children: A randomised controlled trial. Eur J Anaesthesiol. 2019 Oct;36(10):728-737. doi: 10.1097/EJA.0000000000001059. PMID 31356373
- [Background] Garcia De Avila MA, Prata RA, Jacob FLDS, Nobrega FMO, De Barros GR, Sugiura BMG. Educational intervention through a comic book for preoperative anxiety in children, adolescents, and their parents: A randomized clinical trial. J Pediatr Nurs. 2022 Nov-Dec;67:e208-e214. doi: 10.1016/j.pedn.2022.07.010. Epub 2022 Jul 21. PMID 35871148
- [Background] Kalra N, Sabherwal P, Tyagi R, Khatri A, Srivastava S. Relationship between subjective and objective measures of anticipatory anxiety prior to extraction procedures in 8- to 12-year-old children. J Dent Anesth Pain Med. 2021 Apr;21(2):119-128. doi: 10.17245/jdapm.2021.21.2.119. Epub 2021 Mar 31. PMID 33880405
- [Background] Bawaeda O, Wanda D, Aprillia Z. Effectiveness of pop-it therapeutic play on children's anxiety during inhalation therapy in children's wards. Pediatr Med Chir. 2023 Mar 28;45(s1). doi: 10.4081/pmc.2023.315. PMID 36974915
- [Background] Liguori S, Stacchini M, Ciofi D, Olivini N, Bisogni S, Festini F. Effectiveness of an App for Reducing Preoperative Anxiety in Children: A Randomized Clinical Trial. JAMA Pediatr. 2016 Aug 1;170(8):e160533. doi: 10.1001/jamapediatrics.2016.0533. Epub 2016 Aug 1. PMID 27294708
- [Background] Batuman A, Gulec E, Turktan M, Gunes Y, Ozcengiz D. Preoperative informational video reduces preoperative anxiety and postoperative negative behavioral changes in children. Minerva Anestesiol. 2016 May;82(5):534-42. Epub 2015 Oct 16. PMID 26474268
- [Background] Vagnoli L, Bettini A, Amore E, De Masi S, Messeri A. Relaxation-guided imagery reduces perioperative anxiety and pain in children: a randomized study. Eur J Pediatr. 2019 Jun;178(6):913-921. doi: 10.1007/s00431-019-03376-x. Epub 2019 Apr 3. PMID 30944985
- [Background] Kain ZN, Caldwell-Andrews AA, Maranets I, McClain B, Gaal D, Mayes LC, Feng R, Zhang H. Preoperative anxiety and emergence delirium and postoperative maladaptive behaviors. Anesth Analg. 2004 Dec;99(6):1648-1654. doi: 10.1213/01.ANE.0000136471.36680.97. PMID 15562048
- [Background] Kain ZN, Wang SM, Mayes LC, Caramico LA, Hofstadter MB. Distress during the induction of anesthesia and postoperative behavioral outcomes. Anesth Analg. 1999 May;88(5):1042-7. doi: 10.1097/00000539-199905000-00013. PMID 10320165
- [Background] Schober P, Boer C, Schwarte LA. Correlation Coefficients: Appropriate Use and Interpretation. Anesth Analg. 2018 May;126(5):1763-1768. doi: 10.1213/ANE.0000000000002864. PMID 29481436
- [Background] von Baeyer CL, Spagrud LJ. Systematic review of observational (behavioral) measures of pain for children and adolescents aged 3 to 18 years. Pain. 2007 Jan;127(1-2):140-50. doi: 10.1016/j.pain.2006.08.014. Epub 2006 Sep 25. PMID 16996689
- [Background] Goresky GV, Whitsett SF. Psychological preparation of children for surgery. Can J Anaesth. 1994 Nov;41(11):1033-5. doi: 10.1007/BF03015649. No abstract available. English, French. PMID 7828247
- [Background] Kain ZN, Mayes LC, Caramico LA. Preoperative preparation in children: a cross-sectional study. J Clin Anesth. 1996 Sep;8(6):508-14. doi: 10.1016/0952-8180(96)00115-8. PMID 8872693